CLINICAL TRIAL: NCT05712486
Title: Effects on Pain Anda Range of Motion of High Force Lateral Distraction Mobilization of the Hip in Athletes With Hip-related Groin Pain. A Randomized Controlled Trial.
Brief Title: Manual Therapy for the Treatment of Athletic Pubalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Silvia Lahuerta Martín, PH D student, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASVE-NM-22-623
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Osteitis Pubis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double- blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral distraction group (Experimental): High force lateral distraction of affected hip.
  Interventions: Other: High force hip Lateral distraction
- Placebo distraction group (Sham Comparator): Placebo lateral traction of affected hip.
  Interventions: Other: Placebo force hip lateral distraction

INTERVENTIONS:
Other: High force hip Lateral distraction — Hip lateral distraction in adjusted position of maximun flexion and internal rotation, with neutral position of abduction/adduction applying high force of distraction.
  Arms: Lateral distraction group
Other: Placebo force hip lateral distraction — Hip lateral distraction in adjusted position of maximun flexion and internal rotation, with neutral position of abduction/adduction applying placebo force of distraction.
  Arms: Placebo distraction group

SUMMARY:
Athletic osteitis pubis is a high prevalent pathology among athletes, especially in those who make quick change of direction of the movement, like runners or footballers. Despite the fact that there is evidence about conservative treatments, there is a lack of evidence about manual therapy (MT) techniques applied in isolation and its consequences in pain and range of movement. The investigators decided to conduct a randomized controlled trial to compare the effects of a MT technique with placebo technique.

ELIGIBILITY:
Inclusion Criteria:

* Athletes diagnosed with osteitis pubis stage 1 with at least 3 months of evolution.
* Internal rotation ROM limited.
* Positive provocation pain tests.

Exclusion Criteria:

* Pain due to intraarticular hip pathology.
* Hip pain due to inflamatory diseases.
* Previous surgical interventions in hip, pelvis or lumbar spine.
* MRI results or provocation pain tests inconcluyent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Actual PAIN | Baseline
  actual pain reported by the patient using visual analog scale (VAS) from 0 to 10, in which higher scores are worse.
Actual PAIN | after to two weeks of treatment
  actual pain reported by the patient using visual analog scale (VAS)from 0 to 10, in which higher scores are worse.
Actual PAIN | 3 months follow-up
  actual pain reported by the patient using visual analog scale (VAS) from 0 to 10, in which higher scores are worse.
Last week PAIN | Baseline
  past week pain reported by the patient using visual analog scale (VAS) from 0 to 10, in which higher scores are worse.
Last week PAIN | after to two weeks of treatment
  past week pain reported by the patient using visual analog scale (VAS) from 0 to 10, in which higher scores are worse.
Last week PAIN | 3 months follow-up
  past week pain reported by the patient using visual analog scale (VAS) from 0 to 10, in which higher scores are worse.

SECONDARY OUTCOMES:
Range of Movement (ROM) | Baseline
  Hip ROM as described by Pua et al. (2008)
Range of Movement (ROM) | after to two weeks of treatment
  Hip ROM as described by Pua et al. (2008)
Range of Movement (ROM) | 3 months follow-up
  Hip ROM as described by Pua et al. (2008)
Global Rating of Change | after to two weeks of treatment
  Subjective impression as described in GROC scale by Jaeschke, Singer & Guyat (1989)
Global Rating of Change | 3 months follow-up
  Subjective impression as described in GROC scale by Jaeschke, Singer & Guyat (1989)
Group of treatment assignment | after to two weeks of treatment
  Question about which group of treatment was the patient assigned in.
Group of treatment assignment | 3 months follow-up
  Question about which group of treatment was the patient assigned in.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Lahuerta Martín, Principal Investigator — University of Valladolid
Locations (1):
- Silvia Lahuerta Martín, Soria, Spain

IPD SHARING:
Plan to Share IPD: No